CLINICAL TRIAL: NCT04211571
Title: Randomized Controlled Trial of Theranova Versus High-flux Dialyzer on Preservation of REsidual RenAl Function in Incident HemoDialysis Patients (THREAD)
Brief Title: Theranova Versus High-flux Dialyzer on Preservation of Residual Renal Function
Acronym: THREAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: Kyungpook National University Chilgok Hospital (Other); Yeungnam University Hospital (Other); Ewha Womans University (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Yong-Lim Kim, M.D., Ph.D., Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNU-Theranova-01
Record Dates: First submitted 2019-12-21; First posted 2019-12-26 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: End Stage Renal Disease
Keywords: End-stage renal disease; Medium cut-off dialyzer; High-flux dialyzer; Residual renal function
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCO group (Experimental): Hemodialysis using Theranova 400 dialyzer
  Interventions: Device: Theranova 400 dialyzer
- High-flux group (Active Comparator): Hemodialysis using high-flux dialyzer (Fx CorDiax 80; Fresenius Medical Care)
  Interventions: Device: High-flux dialyzer

INTERVENTIONS:
Device: Theranova 400 dialyzer — Hemodialysis using Theranova 400 dialyzer
  Arms: MCO group
Device: High-flux dialyzer — Hemodialysis using high-flux dialyzer
  Other Names: Fx CorDiax 80 dialyzer
  Arms: High-flux group

SUMMARY:
Theranova is a novel medium cut-off dialyzer and has better performance for removal of middle molecules compared to conventional hemodialysis. The study investigates the effect of Theranova dialzyer on preserving residual renal function in the incident hemodialysis pateitns compared to high-flux dialzyer. The primary endpoint is change of glomerular filtration rate, calculated using creatinine and urea clearance. The secondary endpoints are serial changes of glomerular filtration rate and daily urine volume, changes of serum middle molecule concentrations, hospitalization, mortality, and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Incident end-stage renal disease ESRD patient receiving hemodialysis for less than 1 month
* 18 years old and older
* Creatinine clearance of more than 2 ml/min
* Agreement to participate in the clinical study
* Vascular access by arteriovenous fistula/graft

Exclusion Criteria:

* Plan for kidney transplantation within 6 months
* Severe volume overloading state
* Dialysis through permanent catheter
* Any hematologic malignancy or monoclonal gammopathy
* Any malignancy
* Active infectious disease
* HIV infection
* Patient enrolled to another study within 3 month from starting the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2023-09-17 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
Change of glomerular filtration rate | Between baseline and 12 months
  Glomerular filtration rate is calculated as the mean of creatinine and urea clearance adjusted for body surface area. The outcome refers to the mean difference of glomerular filtration rate between baseline and after 12 months.

SECONDARY OUTCOMES:
Change of glomerular filtration rate | 0, 3, 6, 9, 12 months
  Calculated as the mean of creatinine and urea clearance adjusted for body surface area
Change of daily urine volume | 0, 3, 6, 9, 12 months
  Total urine output for 24 hours
Change and reduction ratio of inflammatory marker levels | 0, 12 months
  TNF-alpha, GDF-15, etc.
Change of hs-CRP | 0, 12 months
  hs-CRP
Change of Beta 2-microglobulin | 0, 12 months
  Beta 2-microglobulin
Change of kidney injury markers | 0, 12 months
  NGAL, KIM-1, TIMP-2, IGFBP-7, etc
Change of cystatin-C | 0, 12 months
  Cystatin-C
Change and reduction ratio of Kappa and lambda free light chains | 0, 12 months
  Kappa and lambda free light chains
Hospitalization | Through 12-month study duration
  Frequency, cause, etc.
Mortality | Through 12-month study duration
  Deaths number and causes of death
Patient-reported outcome | 0, 12 months
  Using Kidney Disease Quality of Life Questionnaire-36™ (KDQOL-36™; score ranges from 0 to 100 - higher scores represent better quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook national university chilgok hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirsch AH, Lyko R, Nilsson LG, Beck W, Amdahl M, Lechner P, Schneider A, Wanner C, Rosenkranz AR, Krieter DH. Performance of hemodialysis with novel medium cut-off dialyzers. Nephrol Dial Transplant. 2017 Jan 1;32(1):165-172. doi: 10.1093/ndt/gfw310. PMID 27587605
- [Derived] Lim JH, Seo YJ, Jeon Y, Jeon YH, Jung HY, Choi JY, Park SH, Kim CD, Kang SH, Ryu JH, Kang DH, Cho JH, Kim YL. Expanded Hemodialysis with Theranova Dialyzer and Residual Kidney Function in Patients Starting Long-Term Hemodialysis: A Randomized Controlled Trial. J Am Soc Nephrol. 2025 Mar 4;36(8):1614-1625. doi: 10.1681/ASN.0000000655. PMID 40036081